CLINICAL TRIAL: NCT07082517
Title: Observational Study of Risk Factors for Peripheral Artery Disease in Bathroom Scale Withings Body Cardio Users
Acronym: OBAOMI
Status: Completed | Type: Observational
Sponsor: Withings (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-A02620-39
Record Dates: First submitted 2021-11-15; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: PAD - Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Significant PWV difference: Population with a significant difference PWV between the right and left lower limbs.
  Interventions: Other: Percentage analysis
- No significant PWV difference: Population with no significant difference PWV between the right and left lower limbs.
  Interventions: Other: Percentage analysis

INTERVENTIONS:
Other: Percentage analysis — Analysis the percentage of the population with risk factors that may lead to a PAD.

SUMMARY:
Withings Body Cardio is capable to measure PWV in the right and left lower limbs. The hypothesis of this study is a significant difference in PWV between the right and left lower limbs measured by the device may be the sign of people with more risk factors that may lead to a PAD.

DETAILED DESCRIPTION:
Active users of WITHINGS Body Cardio bathroom scale will be invited to participate to the study. In case of a positive answer, the user will receive an electronic questionnaire about its health and medical history and the data recorded from the previous six months on his/her Body Cardio bathroom scale will be collected in the study.

Once consent has been given, the user's data collectedby the WITHINGS Body Cardio scales will be extracted anonymously and associated with the answers to the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Active and regular user of the device
* Adult participant
* Participant who agreed to participate in the study, after reading the study information letter
* Participant living in France

Exclusion Criteria:

* User who didn't agreed to participate to the study after reading the study information letter

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Active and regular user of the Withings Body Cardio Bathroom Scale
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Analysis of the distribution of risk factors for people with a high People with significant PWV difference will be compared to people with no significant PWV difference | 1 year
  Chi 2 test between the two population

SECONDARY OUTCOMES:
Acceptability of the device | 1 year
  Amount of daily use of the device

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Boutouyrie, Pr, Principal Investigator — Georges Pompidou European Hospital
Locations (1):
- Withings, Issy-les-Moulineaux, Withings, France

IPD SHARING:
Plan to Share IPD: No